CLINICAL TRIAL: NCT02453308
Title: A Multi-centre, Open-label Randomised Trial to Assess the Efficacy, Safety and Tolerability of Triple Artemisinin-based Combination Therapies (TACTs) Com-pared to Artemisinin-based Combination Therapies (ACTs) in Uncomplicated Falciparum Malaria and to Map the Geographical Spread of Artemisinin and Partner Drug Resistance
Brief Title: A Study by the Tracking Resistance to Artemisinin Collaboration (TRAC)
Acronym: TRACII
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BAKMAL1502
Record Dates: First submitted 2015-04-20; First posted 2015-05-25 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Malaria, Falciparum
Keywords: Artemisinin combination Therapies
MeSH Terms: conditions — Malaria, Falciparum | interventions — bis(tetraheptylammonium)tetraiodocyclopentane tellurate(IV)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ACT-arms (Active Comparator): 1.1 Artemether-lumefantrine for 3 days.
  1.2 Dihydroartemisinin-piperaquine for 3 days
  1.3 Artesunate-Mefloquine for 3 days
  Interventions: Drug: ACT
- TACT-arms (Active Comparator): 2.1: Artemether-lumefantrine for 3 days.plus: Amodiaquine for 3 days.
  2.2: Dihydroartemisinin-piperaquine for 3 days. plus: Mefloquine hydrochloride for 3 days.
  2.3 Dihydroartemisinin-piperaquine for 3 days. plus: Mefloquine hydrochloride for 3 days.
  Interventions: Drug: TACT

INTERVENTIONS:
Drug: ACT — 1. Artemether-lumefantrine for 3 days
  2. Dihydroartemisinin-piperaquine for 3 days.
  3. Artesunate-mefloquine for 3 days
  Arms: ACT-arms
Drug: TACT — 1. Artemether-lumefantrine for 3 days plus Amodiaquine for 3 days.
  2. Dihydroartemisinin-piperaquine for 3 days plus Mefloquine hydrochloride for 3 days.
  3. Dihydroartemisinin-piperaquine for 3 days plus Mefloquine hydrochloride for 3 days.
  Arms: TACT-arms

SUMMARY:
This study is an open-label randomised trial comparing standard ACT treatment with matching triple artemisinin-based combination therapies (TACTs), evaluating efficacy in safety and tolerability. The estimated total sample size is 2040 patients from 16 sites in Asia and 1 site in Africa. There are 2 arm study groups that have 2 treatment arms each.

Study group A:

A.1: Artemether-lumefantrine for 3 days. versus: A.2: Artemether-lumefantrine for 3 days plus Amodiaquine for 3 days.

Study group B:

B.1: Dihydroartemisinin-piperaquine for 3 days. versus: B.2: Dihydroartemisinin-piperaquine for 3 days plus Mefloquine hydrochloride for 3 days.

Study group C:

C.1: Artesunate-mefloquine for 3 days versus: C.2: Dihydroartemisinin-piperaquine for 3 days plus Mefloquine hydrochloride for 3 days.

According to the WHO guideline, all patients except for children under the age of 1 year or a weight below 10 kilograms will also be treated with a single dose of low dose primaquine.

DETAILED DESCRIPTION:
In Laos, Myanmar, Bangladesh, India and DRC, the following two combinations will be used:

1. Artemether-lumefantrine combined with amodiaquine (TACT arm) or
2. Artemether-lumefantrine (ACT arm)

In Myanmar and Vietnam the following two combinations will be used:

1. Dihydroartemisinin-piperaquine combined with mefloquine (TACT arm) or
2. Dihydroartemisinin-piperaquine (ACT arm)

In Cambodia and Thailand the following two combinations will be used:

1. Dihydroartemisinin-piperaquine plus Mefloquine hydrochloride (TACT arm) or
2. Artesunate-mefloquine (ACT arm)

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 6 months to 65 years old
* Acute uncomplicated P. falciparum malaria, confirmed by positive blood smear with asexual forms of P. falciparum (or mixed with non-falciparum species)
* Asexual P. falciparum parasitaemia: 5,000 to 200,000/uL, de-termined on a thin or thick blood film (In Cambodia patients with a parasitaemia of 16 to 200,000/uL are eligible. In DRC patients with a parasitaemia of 10,000 to 250,000/ul are eligi-ble)
* Fever defined as >/= 37.5°C tympanic temperature or a history of fever within the last 24 hours
* Written informed consent (by parent/guardian in case of children)
* Willingness and ability of the patients or parents/guardians to comply with the study protocol for the duration of the study

Exclusion Criteria:

* Signs of severe/complicated malaria
* Haematocrit < 25% or Hb < 5 g/dL at screening (DRC: Hct<15% and Hb <5 g/dL due to high prevalence of anemia).
* Acute illness other than malaria requiring treatment
* For females: pregnancy, breast feeding
* Patients who have received artemisinin or a derivative or an artemisinin containing combination therapy (ACT) within the previous 7 days
* Treatment with mefloquine in the 2 months prior to presentation will be an exclusion criteria in the DHA-P+MQ sites
* History of allergy or known contraindication to artemisinins, or to the ACT or TACT to be used at the site e.g. neuropsychiatric disorders will be a contraindication for the use of mefloquine.
* Previous splenectomy
* QTc-interval > 450 milliseconds at moment of presentation
* Documented or claimed history of cardiac conduction problems
* Earlier participation within the TRACII trial or another trial in the previous 3 months.

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1110 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
PCR corrected efficacy defined as adequate clinical and parasitological response (ACPR) | 42 days

SECONDARY OUTCOMES:
Parasite clearance half-life | 42 days
  Parasite clearance half-life assessed by microscopy as primary parameter to de-termine parasite clearance
Parasite reduction rates and ratios at 24 and 48 hours assessed by microscopy | at 24 and 48 hours
Time for parasite count to fall to 50% of initial parasite density | 42 days
Time for parasite count to fall to 90% of initial parasite density | 42 days
Time for parasite count to fall to 99% of initial parasite density | 42 days
Fever clearance time | 42 days
Incidence of adverse events and serious adverse events | 42 days
Incidence of adverse events concerning markers of hepatic toxicity | 42 days
  Total billirubin, ALT, AST and Alkaline Phosphatase will be measured
Incidence of adverse events concerning markersof renal toxicity | 42 days
  Creatinine will be measured
Incidence of prolongation of the QTc-interval | 3 days
  Incidence of prolongation of the Qtc-interval above 500 ms or > 60ms above baseline values
Change in hemoglobin/hematocrit | 42 days
  Change in hemoglobin/hematocrit on day 1 to 7, 14, 21, 28, 35 and 42 according to geographical location and study arm, stratified for G6PD status
Proportion of patients that reports completing a full course of observed TACT or ACT without withdrawal of consent or exclusion from study | 42 days
Prevalence of Kelch13 mutations of known functional significance | 42 days
Prevalence/incidence of other genetic markers of antimalarial drug resistance | 42 days
Genome wide association with in vivo/in vitro sensitivity parasite phenotype | 42 days
Correlation between SNPs measured in dry blood spots and whole genome sequencing in leukocyte depleted blood samples | 42 days
Transcriptomic patterns at t=0 and t=6h comparing sensitive and resistant parasites | 6hrs after start of treatment
Correlation between qPCR based versus microscopy based assessments of parasite clearance dynamics | 14 days
Proportion of patients with gametocytemia before,after treatment with Primaquine | assessed at admission, up to day 14
Levels of RNA transcription coding for male or female specific gametocytes | at admission up to day 14
In vitro sensitivity (expressed in IC50 values among others) of P. falciparum to artemisinins and partner drugs | 42 days
• Pharmacokinetic profiles and interactions of artemisinin-derivatives and partner drugs (half-life, Cmax, AUC, Tmax) in 20 ACT treated and 20 TACT treated patients of both study arms | 42 days
Day 7 drug levels of partner drugs in association with treatment efficacy and treatment arm | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Arjen Dondorp, MD, Principal Investigator — Mahidol Oxford Tropical Medicine Research Unit
Locations (20):
- College of Medicine Chittagong, Rāmu, Bangladesh
- Burma (4):
  - Ann Hospital, Ann Town
  - Pyay hospital, Prome
  - Pyin oo Lwin hospital, Pyin Oo Lwin
  - Thabeikkyin hospital, Thabeikkyin
- Cambodia (4):
  - Pailin, Pailin
  - Preah Vihear, Preah Vihear
  - Pursat, Pursat
  - Ratanakiri, Ratankiri
- Kinshasa, Kinshasa, Democratic Republic of the Congo
- India (3):
  - Ispat General hospital, Rourkela, Rourkela
  - Mohanpur Community health center, Agartala
  - Midnapore, Medinīpur
- Sekong, Sekong, Laos
- Thailand (5):
  - Phusing hospital, Phusing, Changwat Si Sa Ket
  - Tha Song Yang hospital, Tha Song Yang, Changwat Tak
  - Chumphon hospital, Chumphon
  - Kunhan Hospital, Si Sa Ket
  - Thanto Hospital, Yala
- Binh Phuoc hospital, Bình Phước, Vietnam

REFERENCES:
- [Derived] van der Pluijm RW, Tripura R, Hoglund RM, Pyae Phyo A, Lek D, Ul Islam A, Anvikar AR, Satpathi P, Satpathi S, Behera PK, Tripura A, Baidya S, Onyamboko M, Chau NH, Sovann Y, Suon S, Sreng S, Mao S, Oun S, Yen S, Amaratunga C, Chutasmit K, Saelow C, Runcharern R, Kaewmok W, Hoa NT, Thanh NV, Hanboonkunupakarn B, Callery JJ, Mohanty AK, Heaton J, Thant M, Gantait K, Ghosh T, Amato R, Pearson RD, Jacob CG, Goncalves S, Mukaka M, Waithira N, Woodrow CJ, Grobusch MP, van Vugt M, Fairhurst RM, Cheah PY, Peto TJ, von Seidlein L, Dhorda M, Maude RJ, Winterberg M, Thuy-Nhien NT, Kwiatkowski DP, Imwong M, Jittamala P, Lin K, Hlaing TM, Chotivanich K, Huy R, Fanello C, Ashley E, Mayxay M, Newton PN, Hien TT, Valecha N, Smithuis F, Pukrittayakamee S, Faiz A, Miotto O, Tarning J, Day NPJ, White NJ, Dondorp AM; Tracking Resistance to Artemisinin Collaboration. Triple artemisinin-based combination therapies versus artemisinin-based combination therapies for uncomplicated Plasmodium falciparum malaria: a multicentre, open-label, randomised clinical trial. Lancet. 2020 Apr 25;395(10233):1345-1360. doi: 10.1016/S0140-6736(20)30552-3. Epub 2020 Mar 11. PMID 32171078
- [Derived] van der Pluijm RW, Imwong M, Chau NH, Hoa NT, Thuy-Nhien NT, Thanh NV, Jittamala P, Hanboonkunupakarn B, Chutasmit K, Saelow C, Runjarern R, Kaewmok W, Tripura R, Peto TJ, Yok S, Suon S, Sreng S, Mao S, Oun S, Yen S, Amaratunga C, Lek D, Huy R, Dhorda M, Chotivanich K, Ashley EA, Mukaka M, Waithira N, Cheah PY, Maude RJ, Amato R, Pearson RD, Goncalves S, Jacob CG, Hamilton WL, Fairhurst RM, Tarning J, Winterberg M, Kwiatkowski DP, Pukrittayakamee S, Hien TT, Day NP, Miotto O, White NJ, Dondorp AM. Determinants of dihydroartemisinin-piperaquine treatment failure in Plasmodium falciparum malaria in Cambodia, Thailand, and Vietnam: a prospective clinical, pharmacological, and genetic study. Lancet Infect Dis. 2019 Sep;19(9):952-961. doi: 10.1016/S1473-3099(19)30391-3. Epub 2019 Jul 22. PMID 31345710